CLINICAL TRIAL: NCT05314751
Title: Learning to Live With Non-severe Haemophilia
Status: Completed | Type: Observational
Sponsor: Haemnet (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: L2L
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Questionnaire and interview — An online survey and an in-depth interview.

SUMMARY:
While the burden of standard treatment may be reduced through the use of gene therapy, converting those with severe haemophilia to a mild or moderate phenotype, the long-term sequelae of previous joint bleeds and associated limitations imposed on those with severe haemophilia may not translate to lessen the biomedical burden of living with a history of severe haemophilia.

We wish to explore these issues further in the Learning to Live study. The study will also seek to identify the ongoing support needs of those who transition to a milder bleeding phenotype.

DETAILED DESCRIPTION:
Haemophilia is a rare congenital disorder caused by an inherited genetic defect which affects approximately one in every 5,000 males. Haemophilia A (factor VIII [FVIII] deficiency) occurs in 85% of cases with haemophilia B (factor IX [FIX] deficiency) making up the remainder of affected people. Three severities are reported: "severe" (factor activity is less than 1%), "moderate" (factor activity is 1-5% and "mild" (factor activity is 6-25%).

The aim of haemophilia treatment is to reduce the frequency of bleeds, and consequently morbidity and joint damage, in order to prevent future disability. Historically treatment has been replacement of the missing clotting factor when a bleed occurs (on-demand treatment) or regularly and intermittently (prophylactic treatment). With this in developed countries, life expectancy of persons with haemophilia, is expected to be close to normal. Treatment is burdensome for affected individuals and caregivers with treatment complications, (presence of inhibitors, pain, and arthropathy), psychological (stress and coping, anxiety and depression, stigmatisation and discrimination) and economic aspects.

Whilst those with mild haemophilia usually only experience bleeding with trauma or surgery and are less engaged with haemophilia care, the impact of living with mild haemophilia on quality of life is becoming more recognised and further research within this cohort of people is required.

The present day focus of treatment is on normalising individual's lives and reducing treatment burden by using innovative therapies to limit and/or eliminate bleeding episodes. This results in a cohort of individuals who are now living with a less severe phenotype of haemophilia, who may be less able to recognise and treat bleeds and for whom clinical follow up and outcomes will be considerably different to that of their predecessors.

A holistic approach to follow up is required, and should include patient relevant outcome. Living with mild haemophilia is still limiting and when bleeds occur the impact is not mild; many cannot self-infuse, do not recognise when to attend hospital and suffer pain and mobility issues.

This study, which has been co-created with a person with haemophilia, aims to explore the impact of these new treatments using mixed methods study. This includes quantitative data from patient reported outcome assessment (the PROBE validated haemophilia questionnaire) and through in depth qualitative interviews.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of haemophilia A or B of any severity

Exclusion Criteria:

Diagnosis of any other bleeding disorder

Ages: 16 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with haemophilia A or B either mild moderate or severe living in the UK.
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
To Identify and understand the differences between those with genetically mild/moderate haemophilia and those with previously severe haemophilia who have received phenotype altering treatment | 3 months
  Survey using the validated PROBE questionnaire (using 7 point Likert scale)

SECONDARY OUTCOMES:
To assess the impact of phenotype altering treatments on those who receive them, and to compare this with those people with genetically mild/moderate haemophilia. | 3 months
  Interview

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared beyond the study group.